CLINICAL TRIAL: NCT05695222
Title: Comparison of the Prognostic Capacity of Existing Staging Systems for Cutaneous Squamous Cell Carcinoma
Brief Title: Cutaneous Squamous Cell Carcinoma Staging Study
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 291683
Record Dates: First submitted 2022-12-22; First posted 2023-01-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is not an interventional study — This is not an interventional study

SUMMARY:
Cutaneous squamous cell carcinoma (CSCC) is the second most common form of skin cancer, and one of the most common cancers worldwide. The majority of CSCCs are easily removed by surgery and have excellent prognosis. However, a small subset has poor outcomes, including secondary spread in the body (metastasis) and death.

The investigators will look at existing CSCC in people from two UK dermatology centres. The investigators will then evaluate the accuracy of current staging systems in predicting risk of poor outcomes in people. The investigators hope that this project will improve the management of patients with CSCC by validating the predictive power of currently available histological staging classifications for cSCC. In the second stage of the study, The investigators will see whether better prediction tools can be found.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old with diagnosis of CSCC

Exclusion Criteria:

* Patients who decline for their data to be used for research purposes

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated at two tertiary Dermatology centers
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2028-06-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence or metastasis | 4 years
  Proportion of patients developing cutaneous squamous cell carcinoma locoregional recurrence, nodal or distant metastases

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Whipps Cross University Hospital, London
  - Dr Emilia Peleva, London

IPD SHARING:
Plan to Share IPD: No